CLINICAL TRIAL: NCT03789331
Title: Anogenital Distance Differences Between Transgender Males and Female Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Adnan Orhan, Obstetrician and Gynecologist (M.D. and researcher), Uludag University
Other Study IDs: UU-SUAM-2017-21/37
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Sexual Orientation Conflict Disorder
Keywords: transgender males; anogenital distance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transgender Male individuals: * Group Description: This group consists of transgender male individuals who come to the gynecology clinic for medico-legal evaluation before the sex reassignment surgery.
  * Intervention: Anogenital distance measurement with a digital caliper in centimeters in the lithotomy position.
  Interventions: Other: Anogenital distance measurement
- Normal healthy female individuals: * Group Description: Healthy women with normal sexual orientation.
  * Intervention: (The same) Anogenital distance measurement with a digital caliper in centimeters in the lithotomy position.
  Interventions: Other: Anogenital distance measurement

INTERVENTIONS:
Other: Anogenital distance measurement — The women were kindly asked to lay down in the lithotomy position with their thighs at 45° to the examination table. A digital caliper (Mitutoyo 500-752-10 ABSOLUTE Digimatic Coolant Proof Caliper 0-150mm / 0-6", Mitutoyo Corporation, Japan) was used to measure anogenital distance.
  Anogenital distance anus to clitoris: will be measured in centimeters from the anterior clitoral surface to the center of the anus.
  Anogenital distance anus to fourchette: will be measured in centimeters from the posterior fourchette to the center of the anus.
  Two investigators who were blind to the gynecological status of the women will measure each distance three times, and the mean value of the six measurements of each anogenital distance will be used.

SUMMARY:
This study evaluates the anogenital distance measurement differences between transgender male individuals and normal healthy female individuals. Half of the participants will be selected from the men with a masculine gender identity who were assigned female sex at birth (Woman who wanted to be a man). Transgender men will be evaluated with the vaginal examination, and anogenital distance will be measured at the time of gynecological medico-legal evaluation before the sex reassignment surgery. While the other half of the participants will be selected from healthy female individuals, ordinary healthy women will be selected from patients who come to the gynecology clinic for another reason (Women with normal sexual orientation).

DETAILED DESCRIPTION:
There is considerable evidence in human beings and in animal models supporting that anogenital distance as a sensitive biomarker of prenatal androgen reflection of reproductive health and sexual orientation. Anogenital distance is approximately twice as long in male animals compared to female animals, and it is routinely used to determine the natal or birth-assigned sex.

Studies have shown alterations in anogenital distance associated with reproductive health and sexual orientation. For instance, shorter anogenital distance has been reported in boys with hypospadias and cryptorchidism. Men with reduced testicular volume have significantly shorter anogenital distance compared with controls. Increased anogenital distance has been indicated in girls with congenital adrenal hyperplasia.

The investigators hypothesized that a prenatal pathological androgenic environment, resulting in a longer anogenital distance, will be able to be associated with a higher risk of sexual orientation disorders like transsexualism. This cross-sectional study aimed to assess the anogenital distance measurement differences between transgender male persons and normal healthy female individuals.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 18-50 years old.
* Healthy transgender male individuals whose gender identity (Male) are different from their birth-assigned sex (Female). The participants will be invited to the study at the time of medico-legal evaluation before the sex reassignment surgery.

Exclusion Criteria:

* Individuals who are older than 50 (People older than 50 cannot change their gender legally in Turkey).
* Other sexual orientation disorders. (Lesbian, Gay, Bisexual, Queer, Intersex, or Asexual persons)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be healthy transgender male individuals whose gender identity (Male) are different from their birth-assigned sex (Female). These individuals are healthy biologically female persons and want to change their gender to male status. In Turkey, if a woman wants to change her gender, she has to bring a lawsuit against the birth registration office to change her gender to male status. Medico-legal assessments then have to be made at a tertiary gynecological center through the court. The participants will be invited to the study at the time of medico-legal evaluation before the sex reassignment surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-02-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Anogenital Distance (Anus-Clitoris) | 1 hour
  Anogenital Distance (Anus-Clitoris) will be measured from the anterior clitoral surface to the centre of the anus with a digital caliper in centimeters.
Anogenital Distance (Anus-Posterior Fourchette) | 1 hour
  Anogenital Distance (Anus-Posterior Fourchette) will be measured from the posterior fourchette to the centre of the anus with a digital caliper in centimeters.

SECONDARY OUTCOMES:
Anti-Mullerian Hormone (AMH) level measurement | 8 hours
  All blood samples will be collected in the morning after the patient has fasted for at least 8 hours.
FSH (Follicle-stimulating hormone), LH (Luteinizing hormone), Estradiol, and Testosteron level measurements | 8 hours
  All blood samples will be collected in the morning after the patient has fasted for at least 8 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Orhan, M.D., Study Director — Uludag University, Department of Obstetrics and Gynecology
Locations (1):
- Uludag University Hospital, Department of Obstetrics and Gynecology, Bursa, Ozluce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available within 9 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Wu Y, Zhong G, Chen S, Zheng C, Liao D, Xie M. Polycystic ovary syndrome is associated with anogenital distance, a marker of prenatal androgen exposure. Hum Reprod. 2017 Apr 1;32(4):937-943. doi: 10.1093/humrep/dex042. PMID 28333243
- [Background] Sanchez-Ferrer ML, Mendiola J, Hernandez-Penalver AI, Corbalan-Biyang S, Carmona-Barnosi A, Prieto-Sanchez MT, Nieto A, Torres-Cantero AM. Presence of polycystic ovary syndrome is associated with longer anogenital distance in adult Mediterranean women. Hum Reprod. 2017 Nov 1;32(11):2315-2323. doi: 10.1093/humrep/dex274. PMID 29025054